CLINICAL TRIAL: NCT07125820
Title: Effects of Transcutaneous Electrical Nerve stimulatıon and Exercise Training on Pain and functionalıty in Women With Migraine
Brief Title: A Dual Intervention in Migraine Treatment: Tens and Exercise
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Nur ALP, Lecturer, MSc., Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BaskentU-FTR-KA25/136
Record Dates: First submitted 2025-07-25; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Migraine
Keywords: Migraine; Tens; Exercise
MeSH Terms: conditions — Migraine Disorders; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The study is planned as a randomized controlled prospective clinical trial. Study Group In addition to drug treatment and patient education, TENS application and exercise program will be given to the individuals in the study group.Patients will be treated at Isparta Süleyman Demirel University Department of Neurology. The treatment program will last 3 days a week for a total of 8 weeks.
  Control Group Individuals in the control group will receive a single session of placebo TENS application and home exercise program in addition to drug treatment and patient education
Who Masked: Participant
Masking Description: A single-blind study was designed in which the patients would be unaware of their group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patient education, TENS application and Exercise program (Experimental): Study Group In addition to drug treatment and patient education, TENS application and exercise program will be given to the individuals in the study group.Patients will be treated at Isparta Süleyman Demirel University Department of Neurology. The treatment program will last 3 days a week for a total of 8 weeks.In this group, TENS application will be performed 3 days a week, 1 session a day for 8 weeks. Cefar brand digital device of Chattanoga company TENS will be used in the application. The frequency will be set as 100 Hz and the transition time as 100 µsec. The application will be performed for 20 minutes.Patients in this group will be given an exercise program 3 days a week for 8 weeks under the supervision of a physiotherapist. The program will include cervical stabilization exercises, stretching and balance exercises. The program is planned in accordance with the principle of progression from easy to difficult every two weeks and is given in.
  Interventions: Other: Experimental Group
- Placebo TENS Application,Home Exercise Program and patient education program (Active Comparator): Control Group Individuals in the control group will receive a single session of placebo TENS application and home exercise program in addition to drug treatment and patient education.This program will only consist of stretching exercises for the trapezius and levator scapula muscles. The exercises will be recommended to be performed once a day, 3 days a week, for 8 weeks with 10 repetitions. The number, frequency and duration of the exercises will not be increased. The home program will not be followed up by the physiotherapist
  Interventions: Other: control group

INTERVENTIONS:
Other: Experimental Group — There are two groups: a study group and a control group. Both groups will continue taking their doctor-prescribed medications for migraine attacks. After the initial assessment, both groups will receive a 30-minute education and brochure containing lifestyle recommendations to address migraine triggers. The brochure will include recommendations for nutrition, environment, sleep, physical activity, and stress. Additionally, a Chattanooga Cefar® TENS device will be used. The frequency will be set at 100 Hz and the transition time will be set at 100 µs. The session will last 20 minutes. Individuals in the study group will be assigned an exercise program. Patients in this group will exercise in-person three days a week for eight weeks under the supervision of a physical therapist. The program will include cervical stabilization exercises, stretching, and balance exercises. The program is planned with a progression from easy to more difficult every two weeks.
  Arms: Patient education, TENS application and Exercise program
Other: control group — Individuals in the control group will receive a single session of placebo Chattanooga Cefar® TENS application and home exercise program in addition to drug treatment and patient education.Patients in this group will receive a single session of placebo TENS. Electrodes will be placed as in the study group. The physiotherapist will turn on the device but will not increase the current. Thus, the stimulation light of the device will be on but no current will be delivered. Patients will be told that they will not feel anything during the treatment and that this is a feature of the application. The application will be performed for 20 minutes.Home Exercise Program After the initial evaluation and patient education, patients will be offered an exercise program to be performed at home. This program will only consist of stretching exercises for the trapezius and levator scapula muscles. The exercises will be recommended to be performed once a day, 3 days a week, for 8 weeks with 10 repetitions.
  Arms: Placebo TENS Application,Home Exercise Program and patient education program

SUMMARY:
The aim of this clinical trial was to investigate the effects of TENS and exercise training on pain and disability in women diagnosed with migraine. The second aim was to investigate the effects of TENS and exercise training on muscle strength, flexibility, sleep quality, balance, and quality of life in women diagnosed with migraine.

Study hypotheses:

H1: TENS and exercise training are effective on pain in women with migraine. H2: TENS and exercise training are effective on disability in women with migraine.

H3: TENS and exercise training are effective on muscle performance in women with migraine.

H4: TENS and exercise training are effective on flexibility in women with migraine.

H5: TENS and exercise training are effective on sleep quality in women with migraine.

H6: TENS and exercise training are effective on balance in women with migraine. H7: TENS and exercise training are effective on quality of life in women with migraine.

DETAILED DESCRIPTION:
The study will be conducted on volunteer patients diagnosed with migraine by a specialist physician in the Department of Neurology of Isparta Süleyman Demirel University Hospital. All stages of the study will be conducted at Isparta Süleyman Demirel University. Informed consent form will be obtained from all patients participating in the study.

There are two groups in the study: Study and control group. Individuals in both groups will continue the medication recommended by the physician for migraine attacks. In addition, after the initial evaluation, individuals in both groups will be given a session of patient education consisting of lifestyle recommendations for triggering factors in migraine by a specialist physiotherapist, which will last approximately 30 minutes. After this session, patients will be given a brochure prepared by the researchers. The brochure will include recommendations on nutrition, environment, sleep, physical activity and stress Participants.Study Group In addition to drug treatment and patient education, TENS application and exercise program will be given to the individuals in the study group.Patients will be treated at Isparta Süleyman Demirel University Department of Neurology. The treatment program will last 3 days a week for a total of 8 weeks.

Control Group Individuals in the control group will receive a single session of placebo TENS application and home exercise program in addition to drug treatment and patient education.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary female individuals aged 18-55 years
* Being diagnosed with migraine according to the International Headache Society (IHS) criteria
* Having at least 2 migraine attacks per month
* Having started the use of medical medication for migraine treatment 3 months or earlier
* Not taking medication continuously except for migraine attacks

Exclusion Criteria:

* Having vestibular migraine
* Having another type of concomitant headache
* Becoming pregnant
* Being breastfeeding
* History of trauma or surgery in the craniocervical region
* Presence of concomitant neurological (multiple sclerosis, Parkinson's disease, etc.) and/or inflammatory rheumatic diseases (ankylosing spondylitis, rheumatoid arthritis, etc.)
* Presence of psychiatric problems (schizophrenia, bipolar disorder, etc.)
* History of malignancy
* Physiotherapy and rehabilitation for migraine or cervical region in the last 6 months
* Botox / filler application to the face area
* Not attending research sessions regularly or missing 3 consecutive sessions

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-05 (Estimated)

PRIMARY OUTCOMES:
Assessment of Pain | eight weeks and 4th week control after treatment
  Pain intensity, frequency, duration and medication use of the individuals will be evaluated every week with a pain diary. Numeric Pain Scale will be used to assess pain intensity. Individuals will be asked to mark their pain intens
Assessment of Disability | eight weeks
  Migraine Disability Assessment Questionnaire (MIDAS) was developed by Stewart et al. (56) in 1999 to measure migraine-related disability. The Turkish validity and reliability of the scale was studied by Ertaş et al. in 2004 (57). Gedikoğlu et al. (58) demonstrated the validity and reliability of the scale in migraine patients in 2005. The questions in the scale provide the determination of the number of days they cannot participate in school/work, home and leisure time activities due to migraine pain. A total score is obtained with the average score of these five questions. Scoring is divided into 4 groups; Group 1: Little or no impairment (0-5 days missing) Group 2: Mild impairment (6-10 days missing) Group 3: Moderate impairment (11-20 days missing) Group 4: Severe impairment (21 days or more).

SECONDARY OUTCOMES:
Evaluation of Muscle Performance | 8 weeks
  Cranio Cervical Flexion Test will be used to evaluate the performance of the cervical region muscles. "The Stabilizer Pressure Biofeedback Unit" (Chattanoga Group, serial no: 5338276, place of manufacture: U.S) will be used for this test ."It consists of a combined manometer/inflation balloon connected to a pressure cell. In the assessment, the individual will be asked to lie supine on a bed with flexed knees. Then the pressure cell of the instrument will be placed under the suboccipital region without inflating. The manometer will be inflated to 20 mmHg, taking care that the pressure cell does not slip into the lower cervical region. Individuals will be asked to press their chin towards their neck without lifting their head as if saying "yes". They will be asked to repeat this movement 10 times for 10 seconds. The test has 5 stages from 20 mmHg to 30 mmHg. When the patient completes 10 repetitions, the test continues at 22, 24, 26, 28 and 30 mmHg.
Assessing Flexibility | eight weeks
  Back scratch test will be used to assess upper extremity flexibility. In this test, the individual is asked to try to reach the lowest point on his/her back by external rotation of one arm over his/her shoulder with the palm facing his/her back while standing, and to reach the highest point on his/her back by internal rotation of the other arm with the palm facing forward. The distance between the middle fingers of both hands is measured with a tape measure. If the middle fingers do not touch each other, the distance is recorded as "minus" in centimeters, 'zero' if they can reach each other, and "plus" in centimeters if the fingers cross each other
Assessment of Sleep Quality | eight weeks
  The Pittsburgh Sleep Quality Index (PSQI), developed by Buysse et al. (1989), will be used to assess sleep quality. Its Turkish validity and reliability were confirmed by Ağargün et al. The PSQI consists of 24 questions, with 19 self-rated items and 5 answered by a bed partner or roommate (not included in scoring). Of the 19 self-rated questions, 18 are used to calculate the score across seven components: subjective sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. Each component scores 0-3, with a total score range of 0-21. Higher scores indicate poorer sleep quality; scores 0-4 reflect good, and 5-21 poor sleep quality.
Assessing Balance | eight weeks
  The Mini-BESTest, developed by Franchignoni et al. (2010), will be used to assess performance-oriented balance. It is a shortened version of the original BESTest, developed using Rasch analysis. The test includes 14 items grouped into four domains: anticipatory postural adjustments (e.g., sit-to-stand, standing on tiptoes, single-leg stance), reactive postural control (e.g., stepping responses in multiple directions), sensory orientation (e.g., standing on firm/foam/inclined surfaces with eyes open or closed), and dynamic gait (e.g., walking with speed changes, head turns, pivot turns, obstacle navigation, and dual-task walking). Each item is scored on a 3-point scale (0-2), with 0 indicating severe impairment and 2 indicating normal performance. A score of 0 is given if physical assistance is required. The total score ranges from 0 to 28. The Turkish validated version of the Mini-BESTest will be used in the study.
Assessment of Quality of Life | eight weeks
  Headache Impact Test-6 (HIT-6) will be used to evaluate the impact of headache on quality of life (66). The Turkish validity and reliability study of this test was conducted by Dikmen et al. In addition to vitality, pain and psychological distress, areas such as sociability, role and cognitive functioning are evaluated with the HIT-6. While 3 of the 6 items in the test specifically addressed the previous 4 weeks, no specific time interval was specified for the remaining 3 questions. Each item is answered on a 5-point Likert scale (6=never, 8=rarely, 10=sometimes, 11=very often, 13=always). When calculating the total score, the scores of the six items are summed. The total score is between 36 and 78 points. A total score of less than 49 points indicates little or no impact, 50-55 points indicates a little impact, 56-59 points indicates a considerable impact, and 60 points and above indicates a severe impact on quality of life

CONTACTS AND LOCATIONS:
Overall Officials: VEDAT ALİ YÜREKLİ, Neurology Professor, Study Director — Suleyman Demirel University
Locations (1):
- Baskent University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data for the primary and secondary objectives of the research will be compared after they are received.